CLINICAL TRIAL: NCT00463567
Title: A 26-week Treatment, Multicenter, Randomized, Double Blind, Double Dummy, Placebo-controlled, Adaptive, Seamless, Parallel-group Study to Assess the Efficacy, Safety and Tolerability of Two Doses of Indacaterol (Selected From 75, 150, 300 & 600 µg o.d.) in Patients With Chronic Obstructive Pulmonary Disease Using Blinded Formoterol (12 µg b.i.d.) and Open Label Tiotropium (18 µg o.d.) as Active Controls
Brief Title: 26 Week Efficacy, Safety and Tolerability Study of Indacaterol in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: external affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2335S
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Results first posted 2011-08-18 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; COPD; Lung Diseases, Obstructive
Keywords: indacaterol; long acting beta-2 agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — indacaterol; Formoterol Fumarate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (7):
- Indacaterol 150 µg (Continued Into Stage 2) (Experimental): In the morning, Indacaterol 150 µg once daily orally inhaled via a single dose dry powder inhaler (SDDPI) + Placebo to Indacaterol delivered via SDDPI + Placebo to Formoterol delivered via Aerolizer. In the evening, Placebo to Formoterol delivered via Aerolizer. Participated in the 2 week Stage 1 and continued treatment up to 26 weeks in Stage 2. Placebo to Formoterol inhalation in the morning and in the evening was discontinued after Stage 1.
  Daily Inhaled Corticosteroid (ICS) monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Indacaterol; Drug: Placebo to Formoterol
- Indacaterol 300 µg (Continued Into Stage 2) (Experimental): In the morning, Indacaterol 300 µg once daily orally inhaled via a SDDPI + Placebo to Indacaterol delivered via SDDPI + Placebo to Formoterol delivered via Aerolizer. In evening, Placebo to Formoterol delivered via Aerolizer. Participated in the 2 week Stage 1 and continued treatment up to 26 weeks in Stage 2. Placebo to Formoterol inhalation in the morning and in the evening was discontinued after Stage 1.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Indacaterol; Drug: Placebo to Formoterol
- Tiotropium 18 µg (Continued Into Stage 2) (Active Comparator): Tiotropium 18 µg dry powder capsules delivered (open label) via manufacturer's proprietary SDDPI, (Handihaler®). Participated in the 2 week Stage 1 and continued treatment up to 26 weeks in Stage 2.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
  Interventions: Drug: Tiotropium (18 µg o.d.)
- Placebo (Continued Into Stage 2) (Placebo Comparator): In the morning, Placebo to Indacaterol delivered via two SDDPI devices + Placebo to Formoterol delivered via Aerolizer. In the evening, Placebo to Formoterol delivered via Aerolizer. Participated in the 2 week Stage 1 and continued treatment up to 26 weeks in Stage 2. Placebo to Formoterol inhalation in the morning and in the evening was discontinued after Stage 1.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
  Interventions: Drug: Placebo to Indacaterol; Drug: Placebo to Formoterol
- Indacaterol 75 µg (Not Continued into Stage 2) (Experimental): In the morning, Indacaterol 75 µg once daily orally inhaled via a SDDPI + Placebo to Indacaterol delivered via SDDPI + Placebo to Formoterol delivered via Aerolizer. In the evening, Placebo to Formoterol delivered via Aerolizer. Participated in the 2 week Stage 1 but did not continue to Stage 2.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Indacaterol; Drug: Placebo to Formoterol
- Indacaterol 600 µg (Not Continued Into Stage 2) (Experimental): In the morning, 2 capsules of Indacaterol 300 µg once daily orally inhaled via two SDDPI devices + Placebo to Formoterol delivered via Aerolizer. In the evening, Placebo to Formoterol delivered via Aerolizer. Participated in the 2 week Stage 1 but did not continue to Stage 2.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Formoterol
- Formoterol 12 µg (Not Continued Into Stage 2) (Active Comparator): In the morning, Placebo to Indacaterol delivered via two SDDPI devices + Formoterol 12 µg delivered via Aerolizer. In evening, Formoterol 12 µg delivered via Aerolizer. Participated in the 2 week Stage 1 but did not continue to Stage 2.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
  Interventions: Drug: Formoterol (12 µg b.i.d.); Drug: Placebo to Indacaterol

INTERVENTIONS:
Drug: Indacaterol — In the morning, Indacaterol once daily (o.d.) orally inhaled via a single dose dry powder inhaler (SDDPI).
  Arms: Indacaterol 150 µg (Continued Into Stage 2); Indacaterol 300 µg (Continued Into Stage 2); Indacaterol 600 µg (Not Continued Into Stage 2); Indacaterol 75 µg (Not Continued into Stage 2)
Drug: Formoterol (12 µg b.i.d.) — Formoterol 12 µg twice daily (b.i.d.) in the morning and in the evening via an aerolizer.
  Arms: Formoterol 12 µg (Not Continued Into Stage 2)
Drug: Tiotropium (18 µg o.d.) — Tiotropium 18 µg once daily (o.d.) dry powder capsules delivered via a SDDPI.
  Arms: Tiotropium 18 µg (Continued Into Stage 2)
Drug: Placebo to Indacaterol — In the morning, Placebo to Indacaterol once daily (o.d.) orally inhaled via a single dose dry powder inhaler (SDDPI).
  Arms: Formoterol 12 µg (Not Continued Into Stage 2); Indacaterol 150 µg (Continued Into Stage 2); Indacaterol 300 µg (Continued Into Stage 2); Indacaterol 75 µg (Not Continued into Stage 2); Placebo (Continued Into Stage 2)
Drug: Placebo to Formoterol — In the morning and in the evening, placebo to formoterol delivered via Aerolizer.
  Arms: Indacaterol 150 µg (Continued Into Stage 2); Indacaterol 300 µg (Continued Into Stage 2); Indacaterol 600 µg (Not Continued Into Stage 2); Indacaterol 75 µg (Not Continued into Stage 2); Placebo (Continued Into Stage 2)

SUMMARY:
Stage 1 of the study is designed to provide data about the risk-benefit of 4 dose regimens of indacaterol (75, 150, 300 & 600 µg o.d.) in order to select two doses to carry forward into study Stage 2. Study Stage 2 will provide pivotal confirmation of efficacy, safety, and tolerability of the selected indacaterol doses in patients with COPD

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥ 40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure
* Co-operative outpatients with a diagnosis of COPD (moderate to severe as classified by the Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) Guidelines, 2005) and:

  * Smoking history of at least 20 pack years
  * Post-bronchodilator FEV1 < 80% and ≥ 30% of the predicted normal value.
  * Post-bronchodilator FEV1/FVC < 70% (Post refers to within 30 min of inhalation of 400 µg of salbutamol)

Exclusion Criteria:

* Pregnant or lactating females
* Patients who have been hospitalized for a COPD exacerbation in the 6 weeks prior to Visit 1 or during the run-in period
* Patients requiring long term oxygen therapy (> 15 h a day)
* Patients who have had a respiratory tract infection 6 weeks prior to V1 (with further criteria)
* Patients with concomitant pulmonary disease, pulmonary tuberculosis, or clinically significant bronchiectasis
* Patients with a history of asthma (with further criteria)
* Patients with Type I or uncontrolled Type II diabetes
* Patients with contraindications for tiotropium
* Patients who have clinically relevant laboratory abnormalities or a clinically significant abnormality
* Any patient with active cancer or a history of cancer with less than 5 years disease free survival time
* Patients with a history of long QT syndrome or whose QTc interval is prolonged
* Patients with a hypersensitivity to any of the study drugs or drugs with similar chemical structures
* Patients who have had treatment with the investigational drug (with further criteria)
* Patients who have had live attenuated vaccinations within 30 days prior to visit 1, or during run-in period
* Patients with known history of non compliance to medication
* Patients unable to satisfactorily use a dry powder inhaler device or perform spirometry measurements

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2059 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (342):
- United States (219):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pulmonary Medicine Associates PC, Homewood, Alabama
  - Jasper Summit Research, Jasper, Alabama
  - Pulmonary Associate of Mobile, PC, Mobile, Alabama
  - Pulmonary Associates, PA, Glendale, Arizona
  - Pulmonary Associates, PA, Phoenix, Arizona
  - Novartis Investigative Center, Scottsdale, Arizona
  - Arizona Pulmonary Specialists, LTD, Scottsdale, Arizona
  - Premiere Pharmaceutical Research, LLC, Tempe, Arizona
  - Canyon Clinical Research, LLC, Tucson, Arizona
  - SAVAHSC / Pulmonary Section, Tucson, Arizona
  - Novartis Investigator Site, Pine Bluff, Arkansas
  - Novartis Investigator Site, Buena Park, California
  - USC Rancho Amigos Medical Center, Downey, California
  - Encompass Clinical Research - North Coast, Encinitas, California
  - California Research, Fullerton, California
  - Allergy and Asthma Specialists Medical Group and research Center, Huntington Beach, California
  - Interlink Research Institute, Los Alamitos, California
  - Allergy Research Foundation, Inc, Los Angeles, California
  - Novartis Investigator Site, Los Angeles, California
  - Southern California Institute for Respiratory Diseases, Los Angeles, California
  - David Geffen UCLA School of Medicine, Los Angeles, California
  - Advance Clinical Research Institute, Orange, California
  - California Allergy & Asthma Medical Group, Palmdale, California
  - Intergrated Research Group, Riverside, California
  - Allergy & Asthma Associates of Santa Clara Res. Center, San Jose, California
  - Greater Los Angeles Healthcare System, Sepulveda, California
  - Encompass Clinical Research, Spring Valley, California
  - Bensch Clinical Research Associates, Stockton, California
  - Peninsula Pulmonary Medical Associates, Torrance, California
  - Progressive Clinical Research, Vista, California
  - Allergy and Asthma Clinical Research Inc, Walnut Creek, California
  - Boulder Medical Center, Boulder, Colorado
  - National Jewish Medical & Research Center, Denver, Colorado
  - Northern Colorado Pulmonary Consultants, PC, Fort Collins, Colorado
  - New West Physicians Clinical research, Golden, Colorado
  - Rocky Mountain Center for Clinical Research, Wheat Ridge, Colorado
  - Western States Clinical Research, Wheat Ridge, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - Lung Health & Sleep Enhancement Center, Newark, Delaware
  - Clinical Research of West Florida, Clearwater, Florida
  - University of Florida Shands Hospital, Gainesville, Florida
  - Shands Jacksonville Medical Center, Jacksonville, Florida
  - Innovative Research of West Florida, Largo, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Elite Research Institute, Miami, Florida
  - Novartis Investigator Site, Pembroke Pines, Florida
  - Emerald Coast Clinical Research, LLC, Pensacola, Florida
  - Pensacola Research Consultants, Pensacola, Florida
  - Integrity Research, Pensacola, Florida
  - Brevard Pulmonary Specialists, Rockledge, Florida
  - Asthma & Allergy Research Center, Sarasota, Florida
  - South Miami Clinical Research, LLC, South Miami, Florida
  - Central Medical Group, PA, Tamarac, Florida
  - Clireco, Inc, Tamarac, Florida
  - Novartis Investigator Site, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Neutrotrials Research Inc, Atlanta, Georgia
  - Georgia Clinical Research, Austell, Georgia
  - Marietta Pulmonary Medicine, Marietta, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - Southern Illinois Clinical Research Center, O'Fallon, Illinois
  - Novartis Investigator Site, River Forest, Illinois
  - Community Hospital Anderson, Anderson, Indiana
  - Dawes Fretzin Clinical Research Group LLC, Indianapolis, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Iowa Clinical Research Corporation, Iowa City, Iowa
  - University of Iowa, Iowa City, Iowa
  - Heart of America Research Institute, Shawnee Mission, Kansas
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - Novartis Investigator Site, Crescent Springs, Kentucky
  - Kentucky Medical research Center, Lexington, Kentucky
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Family Asthma and Allergy Research Associates, Louisville, Kentucky
  - Gulf Coast Research, LLC, Lafayette, Louisiana
  - Rx R&D, Metaire, Louisiana
  - LSU Health Sciences Center/LSU School of Medicine, New Orleans, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Louisiana Health Sciences Center, Shreveport, Louisiana
  - Northshore Research Associates, Slidell, Louisiana
  - Allergy, Asthma, Immunology, Pharmaceutical Studies, Bangor, Maine
  - Primecare Physician Associates, Biddeford, Maine
  - John Hopkins Asthma and Allergy Center, Baltimore, Maryland
  - Miray Medical Center, Brockton, Massachusetts
  - Fallon Clinic at Worcester Medical Center, Worcester, Massachusetts
  - ClinSite, Inc, Ann Arbor, Michigan
  - Novartis Investigator Site, Clarkston, Michigan
  - Harper University Hospital; Wayne State University, Detroit, Michigan
  - Novartis Investigator Site, Flint, Michigan
  - Pulmonary Respiratory Institute of Southwest Michigan, Livonia, Michigan
  - Novartis Investigator Site, Port Huron, Michigan
  - Synergy Medical Education Alliance, Saginaw, Michigan
  - Novartis Investigator Site, Troy, Michigan
  - Minnesota Lung Center, Edina, Minnesota
  - Clinical Research Institute, Minneapolis, Minnesota
  - Novartis Investigator Site, Minneapolis, Minnesota
  - Minnesota Lung Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Cardio-Pulmonary Research, Chesterfield, Missouri
  - University of Missouri - Columbia, Columbia, Missouri
  - Kansas City University of Medicine and Biosciences, Kansas City, Missouri
  - University of Missouri KC/ Truman Medical, Kansas City, Missouri
  - Midwest Chest Consultants, Saint Charles, Missouri
  - Washington U School of Medicine, Center for Clinical Studies, St Louis, Missouri
  - The Clinical Research Centre, St Louis, Missouri
  - Montana Health Research Institute, Billings, Montana
  - Novartis Investigator Site, Kalispell, Montana
  - Novartis Investigator Site, Missoula, Montana
  - Somnos Laboratories, Inc, Lincoln, Nebraska
  - Omaha VA Medical Center, Omaha, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Midwest Allergy and Asthma Clinic, Omaha, Nebraska
  - Creighton University Centre for Allergy, Asthma & Immunology, Omaha, Nebraska
  - Creigton University, Omaha, Nebraska
  - Heartland Clinical Research, Inc, Omaha, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - University of Nebraska Medical Center - Pulmonary Research, Omaha, Nebraska
  - The Asthma & Allergy Center, PC, Papillion, Nebraska
  - Lovelace Scientific Resources, Inc., Henderson, Nevada
  - Clinical Research Center of NV, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Delaware Valley Clinical Research, Cherry Hill, New Jersey
  - Pulmonary and Critical Care Associates, PA, East Brunswick, New Jersey
  - Novartis Investigator Site, Newark, New Jersey
  - Pulmonary and Allergy Associates, PA, Summit, New Jersey
  - Pulmonary and Critical Care Services, Albany, New York
  - Crescent Medical Associates, Astoria, New York
  - Asthma and Allergy Associates, Cortland, New York
  - Asthma and Allergy Associates, Elmira, New York
  - Nassau Chest Physicians, PC, Massapequa, New York
  - North Shore University Hospital, New Hyde Park, New York
  - New York Pulmonary Associates, PC, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - AAIR research Centre, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Sensenbrenner Primary Care, Charlotte, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Novartis Investigator Site, Shelby, North Carolina
  - Cloverdale Research Facility, Winston-Salem, North Carolina
  - Merit Care Medical Group, Fargo, North Dakota
  - Cincinnati VA Hospital, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Bernstein Clinical Research Centre, Cincinnati, Ohio
  - Community Research Inc, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Metro Health Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University - Davis Heart and Lung Research Institute, Columbus, Ohio
  - Novartis Investigator Site, Columbus, Ohio
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Novartis Investigator Site, Marion, Ohio
  - John Winder Associates, Sylvania, Ohio
  - Advanced Health Care Specialists, Thornville, Ohio
  - The University of Toledo, Toledo, Ohio
  - Pharmacotherapy Research Associates, Inc, Zanesville, Ohio
  - Oklahoma Allergy and Asthma Clinic, Oklahoma City, Oklahoma
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Lynne Health Science Institute, Oklahoma City, Oklahoma
  - Healthcare Research Consultants, Inc, Tulsa, Oklahoma
  - River Road Medical Group, Eugene, Oregon
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Oregon Clinical Research Associates, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Novartis Investigator Site, Portland, Oregon
  - Tri-State Medical Group, Beaver, Pennsylvania
  - Novartis Investigator Site, Easton, Pennsylvania
  - Chest Diseases of Northwestern PA, Erie, Pennsylvania
  - Asthma Allergy &Pulmonary Associates, PC, Philadelphia, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Novartis Investigator Site, Philadelphia, Pennsylvania
  - Pittsburgh Pulmonary Associates, Pittsburgh, Pennsylvania
  - South Hills Pulmonary Associates, Pittsburgh, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Partners in Clinical Research, Cumberland, Rhode Island
  - Low County Lung and Critical Care, PA, Charleston, South Carolina
  - Hugh D. Durrence, MD, Family Medicine, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Med Plus South - Strand Family Practice, Garden City, South Carolina
  - Novartis Investigator Site, Greenville, South Carolina
  - Spartanburg Pharmaceutical Research, Spartanburg, South Carolina
  - Palmetto Pulmonary Medicine, PA - Sleep Disorders Lab, Varnville, South Carolina
  - MultiSpeciality Clinical Research, Johnson City, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Volunteer Research Center, Knoxville, Tennessee
  - Dickson Family Medicine Group, PC, Nashville, Tennessee
  - Novartis Investigator Site, Nashville, Tennessee
  - Heartland Medical, P.C, New Tazewell, Tennessee
  - PharmaTex Research LLC, Amarillo, Texas
  - Trinity Clinic - Corsicana, Corsicana, Texas
  - Pharmaceutical Research & Consulting, Inc, Dallas, Texas
  - Asthma & Allergy Research Associates, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Texas Pulmonary & Critical Care, Fort Worth, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - *Private Practice*, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houstons Veteran's Medical Center, Houston, Texas
  - West Houston Allergy and Asthma, PA, Katy, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Quality Assurance Research Centre, San Antonio, Texas
  - Audie L. Murphy VA Hospital, San Antonio, Texas
  - Allergy and Asthma Research Center, PA, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Wellmed Clinical Research, San Antonio, Texas
  - Vermont Lung Center, Colchester, Vermont
  - Johnston Memorial Hospital Pulmonary Research, Abingdon, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Lynchburg Pulmonary Associates, Lynchburg, Virginia
  - Novartis Investigator Site, Richmond, Virginia
  - Madrona Medical Group - Clinical Research Dept., Bellingham, Washington
  - Pulmonary and Research Associates, Spokane, Washington
  - William L. Gray Research, Spokane, Washington
  - Pulmonary Consultants, PLLC, Tacoma, Washington
  - Madigan Army medical Center / Dept. of Army, Tacoma, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Novartis Investigator Site, Milwaukee, Wisconsin
- Argentina (4):
  - Novartis Investigator Site, Buenos Aires
  - Novartis, Buenos Aires
  - Novartis Investigator Site, Capital Federal
  - Novartis Investigator Site, Santa Fe
- Canada (20):
  - Novartis Investigator Site, Ajax
  - Novartis Investigator Site, Calgary
  - Novartis Investigator Site, Chatham
  - Novartis Investigator Site, Gatineau
  - Novartis Investigator Site, Moncton
  - Novartis Investigator Site, Montreal
  - Novartis Investigator Site, Niagara Falls
  - Novartis Investigator Site, Ottawa
  - Novartis, Québec
  - Novartis Investigator Site, Saint Romuald
  - Novartis Investigator Site, Saskatoon
  - Novartis Investigator Site, Sherbrooke
  - Novartis Investigator Site, St. John's
  - Novartis Investigator Site, Ste-Foy
  - Novartis Investigator Site, Toronto
  - Novartis Investigator Site, Trois-Rivières
  - Novartis Investigator Site, Vancouver
  - Novartis Investigator Site, Waterloo
  - Novartis Investigator Site, Windsor
  - Novartis Investigator Site, Winnipeg
- Germany (21):
  - Novartis Investigator Site, Augsburg
  - Novartis Investigator Site, Bad Segeberg
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Bielefeld
  - Novartis Investigator Site, Bonn
  - Novartis Investigator Site, Brühl
  - Novartis Investigator Site, Dachau
  - Novartis, Fürth
  - Novartis Investigator Site, Hamburg
  - Novartis Investigator Site, Hoyerswerda
  - Novartis Investigator Site, Kaufbeuren
  - Novartis Investigator Site, Landsberg
  - Novartis Investigator Site, Leipzig
  - Novartis Investigator Site, Mainz
  - Novartis Investigator Site, München
  - Novartis Investigator Site, Oranienburg
  - Novartis Investigator Site, Oschersleben
  - Novartis Investigator Site, Potsdam
  - Novartis Investigator Site, Ratingen
  - Novartis Investigator Site, Steinfurt
  - Novartis Investigator Site, Wuppertal
- India (12):
  - Novartis Investigator Site, Bangalore
  - Novartis Investigator Site, Banglore
  - Novartis Investigator Site, Caranazalem
  - Novartis Investigator Site, Chennai
  - Novartis Investigator Site, Coimbatore
  - Novartis Investigator Site, Hyderabaad
  - Novartis Investigator Site, Indore
  - Novartis Investigator Site, Jaipur
  - Novartis Investigator Site, Kolkata
  - Novartis Investigator Site, Ludhiana
  - Novartis Investigator Site, Mumbai
  - Novartis Investigator Site, Trivandrum
- Italy (16):
  - Novartis Investigator Site, Bologna
  - Novartis Investigator Site, Busto Arsizio
  - Novartis Investigator Site, Catania
  - Novartis Investigator Site, Catanzaro
  - Novartis Investigator Site, Chioggia
  - Novartis Investigator Site, Crema
  - Novartis Investigator Site, Ferrara
  - Novartis Investigator Site, Florence
  - Novartis Investigator Site, Genova
  - Novartis Investigator Site, Messina
  - Novartis Investigator Site, Milan
  - Novartis, Milan
  - Novartis Investigator Site, Pisa
  - Novartis Investigator Site, Roma
  - Novartis Investigator Site, Rozzano
  - Novartis Investigator Site, Siena
- Novartis Investigator Site, Ponce, Puerto Rico
- South Korea (9):
  - Novartis Investigator Site, Bucheon-si
  - Novartis Investigator Site, Busan
  - Novartis Investigator Site, Chuncheon
  - Novartis Investigator Site, Daegu
  - Novartis Investigator Site, Kwangju
  - Novartis Investigator Site, Seoul
  - Novartis, Seoul
  - Novartis Investigator Site, Suwon
  - Novartis Investigator Site, Wŏnju
- Spain (23):
  - Novartis Investigator Site, A Coruña
  - Novartis Investigator Site, Alicante
  - Novartis Investigator Site, Barcelona
  - Novartis, Barcelona
  - Novartis Investigator Site, Burgos
  - Novartis Investigator Site, Cadiz
  - Novartis Investigator Site, Calde Lugo
  - Novartis Investigator Site, Galdakano
  - Novartis Investigator Site, Girona
  - Novartis Investigator Site, Gran Canaria
  - Novartis Investigator Site, Madrid
  - Novartis Investigator Site, Málaga
  - Novartis Investigator Site, Ourense
  - Novartis Investigator Site, Oviedo
  - Novartis Investigator Site, Palma de Mallorca
  - Novartis Investigator Site, Ponferrada
  - Novartis Investigator Site, Pontevedra
  - Novartis Investigator Site, Port de Sagunt
  - Novartis Investigator Site, Seville
  - Novartis Investigator Site, Valencia
  - Novartis Investigator Site, Vic
  - Novartis Investigator Site, Vila-real
  - Novartis Investigator Site, Zaragoza
- Sweden (5):
  - Novartis, Gothenburg
  - Novartis Investigator Site, Jönköping
  - Novartis Investigator Site, Lidingö
  - Novartis Investigator Site, Luleå
  - Novartis Investigator Site, Lund
- Taiwan (5):
  - Novartis Investigator Site, Chiayi City
  - Novartis Investigator Site, Linkou District
  - Novartis Investigator Site, Taichung
  - Novartis Investigator Site, Taipei
  - Novartis, Taipei
- Turkey (Türkiye) (7):
  - Novartis Investigator Site, Ankara
  - Novartis, Istanbul
  - Novartis Investigator Site, Izmir
  - Novartis Investigator Site, Konya
  - Novartis Investigator Site, Manisa
  - Novartis Investigator Site, Mersin
  - Novartis Investigator Site, Yenişehir

REFERENCES:
- [Derived] Jones PW, Donohue JF, Nedelman J, Pascoe S, Pinault G, Lassen C. Correlating changes in lung function with patient outcomes in chronic obstructive pulmonary disease: a pooled analysis. Respir Res. 2011 Dec 29;12(1):161. doi: 10.1186/1465-9921-12-161. PMID 22206353
- [Derived] Yelensky R, Li Y, Lewitzky S, Leroy E, Hurwitz C, Rodman D, Trifilieff A, Paulding CA. A pharmacogenetic study of ADRB2 polymorphisms and indacaterol response in COPD patients. Pharmacogenomics J. 2012 Dec;12(6):484-8. doi: 10.1038/tpj.2011.54. Epub 2011 Dec 13. PMID 22158330
- [Derived] Jones PW, Mahler DA, Gale R, Owen R, Kramer B. Profiling the effects of indacaterol on dyspnoea and health status in patients with COPD. Respir Med. 2011 Jun;105(6):892-9. doi: 10.1016/j.rmed.2011.02.013. Epub 2011 Mar 11. PMID 21397482
- [Derived] Worth H, Chung KF, Felser JM, Hu H, Rueegg P. Cardio- and cerebrovascular safety of indacaterol vs formoterol, salmeterol, tiotropium and placebo in COPD. Respir Med. 2011 Apr;105(4):571-9. doi: 10.1016/j.rmed.2010.11.027. Epub 2011 Jan 11. PMID 21227674
- [Derived] Donohue JF, Fogarty C, Lotvall J, Mahler DA, Worth H, Yorgancioglu A, Iqbal A, Swales J, Owen R, Higgins M, Kramer B; INHANCE Study Investigators. Once-daily bronchodilators for chronic obstructive pulmonary disease: indacaterol versus tiotropium. Am J Respir Crit Care Med. 2010 Jul 15;182(2):155-62. doi: 10.1164/rccm.200910-1500OC. Epub 2010 May 12. PMID 20463178

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of two stages: a dose selection stage (Stage 1, 2 weeks) from which 2 out of 4 Indacaterol doses were selected following interim analysis to continue into Stage 2 for comparisons of efficacy, safety, and tolerability for total treatment of up to 26 weeks.
Groups:
- Tiotropium (Continued Into Stage 2): Tiotropium 18 µg dry powder capsules delivered (open label) via manufacturer's proprietary SDDPI, (Handihaler®). Participated in the 2 week Stage 1 and continued treatment up to 26 weeks in Stage 2.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
Period: Overall Study
Arm/Group | Indacaterol 150 µg (Continued Into Stage 2) | Indacaterol 300 µg (Continued Into Stage 2) | Tiotropium (Continued Into Stage 2) | Placebo (Continued Into Stage 2) | Indacaterol 75 µg (Not Continued Into Stage 2) | Indacaterol 600 µg (Not Continued Into Stage 2) | Formoterol 12 µg (Not Continued Into Stage 2)
Started | 420 (Randomized Participants) | 418 | 420 | 425 | 130 | 123 | 123
Safety Population: Received Study Drug | 416 | 416 | 415 | 418 | 127 ('Completed' indicates the number of patients in the interim analysis.) | 122 ('Completed' indicates the number of patients in the interim analysis.) | 122 ('Completed' indicates the number of patients in the interim analysis.)
Completed | 325 | 341 | 331 | 294 | 107 | 102 | 112
Not Completed | 95 | 77 | 89 | 131 | 23 | 21 | 11
Not completed — Adverse Event | 29 | 26 | 17 | 46 | 10 | 10 | 4
Not completed — Withdrawal by Subject | 29 | 22 | 20 | 37 | 6 | 5 | 1
Not completed — Protocol Deviation | 13 | 9 | 14 | 11 | 1 | 1 | 2
Not completed — Lost to Follow-up | 12 | 6 | 13 | 8 | 1 | 1 | 1
Not completed — Administrative problems | 5 | 3 | 6 | 9 | 3 | 2 | 2
Not completed — Lack of Efficacy | 4 | 9 | 9 | 17 | 1 | 0 | 1
Not completed — Abnormal lab value(s) | 1 | 1 | 2 | 1 | 1 | 0 | 0
Not completed — Abnormal test procedure result(s) | 1 | 1 | 6 | 2 | 0 | 2 | 0
Not completed — Death | 1 | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 150 µg (Continued Into Stage 2) | Indacaterol 300 µg (Continued Into Stage 2) | Tiotropium 18 µg (Continued Into Stage 2) | Placebo (Continued Into Stage 2) | Indacaterol 75 µg (Not Continued Into Stage 2) | Indacaterol 600 µg (Not Continued Into Stage 2) | Formoterol 12 µg (Not Continued Into Stage 2) | Total
Number analyzed (Participants) | 416 | 416 | 415 | 418 | 127 | 122 | 122 | 2036
Age, Customized [Number; unit: participants] — Baseline Measures were based on the Safety Population that included all participants who received at least one dose of study drug.
  participants
    Between 40 and 64 years | 214 | 230 | 215 | 215 | 58 | 60 | 56 | 1048
    ≥65 years | 202 | 186 | 200 | 203 | 69 | 62 | 66 | 988
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 153 | 146 | 163 | 51 | 48 | 52 | 770
  Male | 259 | 263 | 269 | 255 | 76 | 74 | 70 | 1266

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) Assessed by Spirometry 24 Hour Post Dose After 12 Weeks of Treatment
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of the 23 h 10 min and the 23 h 45 min post dose values. Mixed model used baseline FEV1, FEV1 prior to and 30 minutes post inhalation of salbutamol/albuterol, and FEV1 prior to and 1 hour post inhalation of ipratropium as covariates.
Time Frame: after 12 weeks of treatment
Population: Participants from the Intent to Treat Population of Stage 2 of the study who received at least one dose of study drug and for whom data was available for FEV1 at 12 weeks. Imputed with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 µg (Continued Into Stage 2) | Indacaterol 300 µg (Continued Into Stage 2) | Tiotropium 18 µg (Continued Into Stage 2) | Placebo (Continued Into Stage 2)
Number analyzed (Participants) | 389 | 389 | 393 | 376
Liters | 1.46 (0.015) | 1.46 (0.015) | 1.42 (0.015) | 1.28 (0.015)

2. Secondary Outcome: The Percentage of "Days of Poor Control" Reported Over the 26 Week Treatment Period
Description: A Chronic Obstructive Pulmonary Disease (COPD) "day of poor control" was defined as any day in the participant's diary with a score ≥2 (moderate or severe) for at least 2 of 5 symptoms (cough, wheeze, production of sputum, color of sputum, breathlessness). Score for each symptom ranges from 0-3; a higher number indicates a more severe symptom. The model contained baseline percentage of "days of poor control" as well as FEV1 reversibility components as covariates.
Time Frame: up to 26 weeks
Population: Intent to Treat population consisting of all participants in Stage 2 of the study who received at least one dose of study drug. Eligible participants for the analysis were those with ≥7 evaluable diary days in the baseline period and ≥30% evaluable diary days (at least 20 days) in total.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Indacaterol 150 µg (Continued Into Stage 2) | Indacaterol 300 µg (Continued Into Stage 2) | Tiotropium (Continued Into Stage 2) | Placebo (Continued Into Stage 2)
Number analyzed (Participants) | 385 | 384 | 391 | 362
Percentage of days | 31.5 (1.51) | 30.8 (1.51) | 31.0 (1.50) | 34.0 (1.53)

3. Other Pre Specified Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) Assessed by Spirometry 24 Hour Post Dose After 2 Weeks of Treatment
Description: Interim Analysis: Stage 1.
  Spirometry was conducted according to internationally accepted standards. Trough FEV1 was defined as the average of the 23 h 10 min and the 23 h 45 min post dose values. Mixed model used baseline FEV1, FEV1 prior to and 30 minutes post inhalation of salbutamol/albuterol, and FEV1 prior to and 1 hour post inhalation of ipratropium as covariates.
Time Frame: Day 15, After 2 Weeks of treatment in Stage 1
Population: Interim Intent-to-treat (ITT) population included participants in Stage 1 of the study who received at least one dose of study drug and for whom data were available for Trough FEV1 at Day 15. Missing data were imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Indacaterol 150 µg: In the morning, Indacaterol 150 µg once daily orally inhaled via a SDDPI + Placebo to Indacaterol delivered via SDDPI + Placebo to Formoterol delivered via Aerolizer. In the evening, Placebo to Formoterol delivered via Aerolizer.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
- Indacaterol 300 µg: In the morning, Indacaterol 300 µg once daily orally inhaled via a SDDPI + Placebo to Indacaterol delivered via SDDPI + Placebo to Formoterol delivered via Aerolizer. In evening, Placebo to Formoterol delivered via Aerolizer.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
- Tiotropium 18 µg: Tiotropium 18 µg dry powder capsules delivered (open label) via manufacturer's proprietary SDDPI, (Handihaler®).
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
- Placebo: In the morning, Placebo to Indacaterol delivered via two SDDPI devices + Placebo to Formoterol delivered via Aerolizer. In evening, Placebo to Formoterol delivered via Aerolizer.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
- Indacaterol 75 µg: In the morning, Indacaterol 75 µg once daily orally inhaled via a SDDPI + Placebo to Indacaterol delivered via SDDPI + Placebo to Formoterol delivered via Aerolizer. In the evening, Placebo to Formoterol delivered via Aerolizer.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
- Indacaterol 600 µg: In the morning, 2 capsules of Indacaterol 300 µg once daily orally inhaled via two SDDPI devices + Placebo to Formoterol delivered via Aerolizer. In the evening, Placebo to Formoterol delivered via Aerolizer.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
- Formoterol 12 µg: In the morning, Placebo to Indacaterol delivered via two SDDPI devices + Formoterol 12 µg delivered via Aerolizer. In evening, Formoterol 12 µg delivered via Aerolizer.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Tiotropium 18 µg | Placebo | Indacaterol 75 µg | Indacaterol 600 µg | Formoterol 12 µg
Number analyzed (Participants) | 105 | 110 | 112 | 104 | 104 | 108 | 105
Liters | 1.49 (0.024) | 1.52 (0.024) | 1.45 (0.023) | 1.31 (0.024) | 1.46 (0.024) | 1.51 (0.024) | 1.42 (0.024)

4. Other Pre Specified Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Time) Area Under the Curve (AUC) From 1 Hour to 4 Hour Post Morning Dose After 2 Weeks of Treatment
Description: Interim Analysis: Stage 1.
  Spirometry was conducted according to internationally accepted standards. Standardized with respect to time (AUC 1h-4h) for FEV1 measurements taken from 1 hour to 4 hour post morning dose on Day 14. Standardized FEV1 AUC was calculated by the trapezoidal rule. Mixed model used baseline FEV1, FEV1 prior to and 30 minutes post inhalation of salbutamol/albuterol, and FEV1 prior to and 1 hour post inhalation of ipratropium as covariates.
Time Frame: Day 14, After 2 Weeks of treatment in Stage 1
Population: Interim Intent-to-treat (ITT) population included participants in Stage 1 of the study who received at least one dose of study drug and for whom data were available for AUC 1h-4h FEV1 at Day 14. Missing data were imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Formoterol 12 µg: In the morning, Placebo to Indacaterol delivered via SDDPI devices + Formoterol 12 µg delivered via Aerolizer. In evening, Formoterol 12 µg delivered via Aerolizer.
  Daily ICS monotherapy (if applicable) was to remain stable and Salbutamol/albuterol was available for rescue use throughout study.
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Tiotropium 18 µg | Placebo | Indacaterol 75 µg | Indacaterol 600 µg | Formoterol 12 µg
Number analyzed (Participants) | 96 | 99 | 99 | 90 | 95 | 97 | 93
Liters | 1.53 (0.034) | 1.58 (0.034) | 1.49 (0.034) | 1.30 (0.033) | 1.50 (0.034) | 1.53 (0.034) | 1.52 (0.035)

ADVERSE EVENTS:
Description: Safety Population including all participants who received at least one dose of study drug.
Arm/Group | Indacaterol 150 µg (Continued Into Stage 2) | Indacaterol 300 µg (Continued Into Stage 2) | Tiotropium 18 µg (Continued Into Stage 2) | Placebo (Continued Into Stage 2) | Indacaterol 75 µg (Not Continued Into Stage 2) | Indacaterol 600 µg (Not Continued Into Stage 2) | Formoterol 12 µg (Not Continued Into Stage 2)
Serious Adverse Events (participants affected / at risk) | 35/416 | 32/416 | 34/415 | 35/418 | 9/127 | 5/122 | 4/122
Other Adverse Events (participants affected / at risk) | 159/416 | 159/416 | 156/415 | 155/418 | 39/127 | 44/122 | 31/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 µg (Continued Into Stage 2) (N=416) | Indacaterol 300 µg (Continued Into Stage 2) (N=416) | Tiotropium 18 µg (Continued Into Stage 2) (N=415) | Placebo (Continued Into Stage 2) (N=418) | Indacaterol 75 µg (Not Continued Into Stage 2) (N=127) | Indacaterol 600 µg (Not Continued Into Stage 2) (N=122) | Formoterol 12 µg (Not Continued Into Stage 2) (N=122)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 1 | 0 | 1 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 3 | 2 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Endocardial fibroelastosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 1 | 3 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster oticus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Mycobacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 4 | 4 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device failure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Glasgow coma scale abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual midline shift syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic peritoneal adhesions (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 | 7 | 7 | 10 | 3 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 3 | 1 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardioversion (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 µg (Continued Into Stage 2) (N=416) | Indacaterol 300 µg (Continued Into Stage 2) (N=416) | Tiotropium 18 µg (Continued Into Stage 2) (N=415) | Placebo (Continued Into Stage 2) (N=418) | Indacaterol 75 µg (Not Continued Into Stage 2) (N=127) | Indacaterol 600 µg (Not Continued Into Stage 2) (N=122) | Formoterol 12 µg (Not Continued Into Stage 2) (N=122)
Bronchitis (Infections and infestations) | 7 | 17 | 13 | 24 | 2 | 3 | 3
Nasopharyngitis (Infections and infestations) | 33 | 39 | 36 | 36 | 7 | 8 | 4
Upper respiratory tract infection (Infections and infestations) | 34 | 27 | 31 | 31 | 10 | 11 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 13 | 6 | 4 | 1 | 9 | 4
Headache (Nervous system disorders) | 28 | 18 | 19 | 14 | 10 | 3 | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 67 | 72 | 75 | 86 | 11 | 19 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 30 | 26 | 27 | 7 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.